CLINICAL TRIAL: NCT06031168
Title: Evaluation the Effect of Topically Coated Dental Implants With 1% Metformin Gel on Osteointegration and Crestal Marginal Bone Loss (a Randomized Controlled Clinical Trial)
Brief Title: 1% Metformin Gel-coated Implants and Osteointegration and Crestal Marginal Bone Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Implants_2023
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Osteointegration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: Metformin gel coated implants
- Control group (Active Comparator)
  Interventions: Other: uncoated hydrophilic dental implants

INTERVENTIONS:
Other: Metformin gel coated implants — Patients will be treated with 1% concentrated metformin gel coated hydrophilic dental implant.
  Arms: Test group
Other: uncoated hydrophilic dental implants — Patients treated by uncoated implants
  Arms: Control group

SUMMARY:
Achieving and maintaining a long term osseointegrated dental implant is a golden goal of success in field of dentistry. Osteointegration depends on surface treatment of dental implants. various techniques of implant coating have been introduced to enhance and accelerate osteointegration. The purpose of present study is to clinically and radiographically evaluate the osseointegration around hydrophilic dental implants coated with 1% Metformin gel Materials and Methods: We executed a randomized controlled clinical trial. The sample will include patients demanding dental implant treatment. Patients will be randomly allocated into the two groups of the study. The group A will be treated with 1% concentrated metformin gel coated hydrophilic dental implant. Group B will be treated with uncoated hydrophilic dental implant. The primary outcome variable will be implant osteointegration and crestal marginal bone loss around implants. It will be measured at time of implant placement and reevaluated after 4, 6-months with periapical x-ray and 3-dimensional imaging.

ELIGIBILITY:
Inclusion Criteria:

* Good general periodontal health and maintenance.
* Adequate amount of bone volume at implant site, allowing to perform the dental implant surgery procedure without bone grafting techniques

Exclusion criteria

* Heavy smokers who smoke more than ten cigarettes per day
* Diabetic patients who have received metformin as antidiabetic drug
* local or systemic conditions that will interfere with routine implant placement (uncontrolled diabetes mellitus or human immune deficiency virus infections, resonance therapy), bone disorders (hyperparathyroidism, osteoporosis, or Paget's disease
* Patients who had subjected to intravenous and/or oral bisphosphonate therapy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-09-04 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in implant stability | Baseline and 4 months
  stability will be assessed by using ostell device

SECONDARY OUTCOMES:
change in marginal bone loss | Baseline and 4 months
  To evaluate the amount of bone loss around osseointegrated implants all patient will be subjected to periapical x-ray.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt